CLINICAL TRIAL: NCT02695992
Title: Rate Control in Atrial Fibrillation II
Acronym: RATAFII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asker & Baerum Hospital (Other)
Collaborators: Vestre Viken Hospital Trust (Other); Helse Sor-Ost (Other Government)
Responsible Party: Principal Investigator, Sara Reinvik Ulimoen, MD PhD postdoc fellow, Asker & Baerum Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 240415; 2015-001918-98 (EudraCT Number)
Record Dates: First submitted 2015-04-28; First posted 2016-03-02 (Estimated); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Atrial Fibrillation; Permanent Atrial Fibrillation
Keywords: Rate control in atrial fibrillation; Beta blockers; Calcium channel blockers; Permanent atrial fibrillation; Management of atrial fibrillation; Atrial fibrillation and biomarkers; Arrhythmias, cardiac; Heart Diseases; Pathological processes; Diltiazem; Metoprolol; Adrenergic Agents; Adrenergic Antagonists; Adrenergic beta-1 Receptor Antagonists; Adrenergic beta-Antagonists; Anti-Arrhythmia Agents; Antihypertensive Agents; Autonomic Agents; Cardiovascular Agents; Membrane Transport Modulators; Molecular Mechanisms of Pharmacological Action; Neurotransmitter Agents; Peripheral Nervous System Agents; Physiological Effects of Drugs; Sympatholytics; Therapeutic Uses; Vasodilator Agents; Troponins; NT-proBNP; Biomarkers
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases; Pathologic Processes | interventions — Metoprolol; Diltiazem

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metoprolol (Active Comparator): Metoprolol, extended release tablets. 100 mg daily
  Interventions: Drug: Metoprolol
- Diltiazem (Active Comparator): Diltiazem, extended release tablets. 360 mg daily
  Interventions: Drug: Diltiazem

INTERVENTIONS:
Drug: Metoprolol — Dosage 100 mg o.d.
  Other Names: Selo-Zok Metoprolol Astra Zeneca depot
  Arms: Metoprolol
Drug: Diltiazem — Dosage 360 mg o.d.
  Other Names: Cardizem Diltiazem Uno depot
  Arms: Diltiazem

SUMMARY:
The RATAF II study is a randomized, prospective, parallel group study, designed to compare the effects of two different drug regimens for rate control in permanent AF (atrial fibrillation). We will investigate on the difference in effects on exercise capacity, biomarkers (NT-proBNP (N-terminal pro-brain natriuretic peptide), troponins, hs-CRP), heart rate, echocardiographic measurements and symptoms.

Our main hypothesis is that six months' treatment with the calcium channel blocker diltiazem will lower NT-proBNP and increase exercise capacity (peak VO2) compared to treatment with the beta blocker metoprolol in permanent AF.

DETAILED DESCRIPTION:
Atrial fibrillation is a common cardiac disease, with increasing incidence and prevalence. There are two main treatment strategies for this arrhythmia, rhythm control and rate control. As rate control is easier to achieve and no major difference in outcome has been found between these two strategies, it is considered a reasonable initial treatment for the majority of AF patients.

Reduced exercise capacity is the most prevalent symptom in patients with permanent AF. In the first Rate control in Atrial Fibrillation (RATAF) study, we demonstrated that calcium channel blockers preserved exercise capacity, reduced arrhythmia-related symptoms and lowered levels of NT-proBNP - whereas the beta blockers reduced the exercise capacity, did not reduce arrhythmia-related symptoms and increased NT-proBNP.

These findings are relevant to a large proportion of patients with permanent AF, suggesting that calcium channel blockers should be the first drug of choice for rate control in patients without heart failure or coronary heart disease. Our results challenge the current widespread use of beta blockers in this setting. However, as the follow up time in the RATAF study was only 3 weeks, it is not clear if these effects are sustained over time. Furthermore, we do not know the mechanisms for the differential effects on exercise capacity, arrhythmia related symptoms and NT-proBNP levels.

In the RATAF II study we will investigate whether the effects on NT-proBNP levels, exercise capacity and symptoms are sustained over time, and explore potential mechanisms that may explain the difference in these effects. The study will provide new insights and results relevant for everyday clinical practice and be of importance for a large and growing group of patients.

A total of 240 patients will be included. Eligible patients will be recruited from the out-patient clinics at the participation hospitals and through advertisements in local newspapers. After inclusion and a wash-out period of 14 days free from drugs affecting the heart rate, patients will be examined by echocardiography, 12-lead ECG (electrocardiography), 24h Holter monitoring, maximal cardiopulmonary exercise test and venous blood sampling at rest, at maximal exercise and after recovery. Perceived arrhythmia related symptoms, quality of life and level of physical activity will be assessed using self-administered questionnaires.

Participants will be randomized through a computer-generated randomization list, to receive one of the study drug regimens; metoprolol 100 mg o.d. or diltiazem 360 mg o.d. The investigators and study personnel will be blinded with regard to allocated study drug. The participants themselves will know what study drug they are assigned. Also, study personnel not involved in examinations will also be able to acquire knowledge concerning assigned study drug, to ensure the process of dosage in the startup phase, assess adverse events (AE) and side effects throughout the study.

Examinations will be repeated after four weeks and six months. All examinations will be performed at the Department of Medical Research, Baerum Hospital to ensure standardized procedures.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age
* Symptomatic, permanent AF of at least three months duration
* Resting heart rate ≥80 bpm
* Signed informed consent

Exclusion Criteria:

* Congestive heart failure
* Ischemic heart disease
* Hypotension (Systolic blood pressure <100 mmHg)
* Treatment with class I or III antiarrhythmic drugs
* Severe hepatic or renal failure
* Pregnancy or lactation
* Hypersensitivity or contradictions to study drugs
* Atrio-ventricular conduction disturbances
* Thyrotoxicosis
* Life limiting disease or substance abuse which may affect participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-02; Primary Completion 2021-10 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Levels of NT-proBNP | 4 weeks
  Levels of NT-proBNP will be measured at baseline and after 4 weeks to assess change
Levels of NT-proBNP | 6 months
  Levels of NT-proBNP will be measured after 6 months

SECONDARY OUTCOMES:
Exercise capacity defined as peak VO2 | 4 weeks
  Exercise capacity will be assessed by cardiopulmonary exercise test at baseline and after 4 weeks to assess change
Exercise capacity defined as peak VO2 | 6 months
  Exercise capacity will be assessed by cardiopulmonary exercise test after 6 months
Ventricular heart rate | 4 weeks
  Ventricular heart rate will be assessed by ECG at rest and during exercise. Will be measured at baseline and after 4 weeks to assess change
Ventricular heart rate | 6 months
  Ventricular heart rate will be assessed by ECG at rest and during exercise. Will be measured after 6 months.
Other biomarkers | 4 weeks
  Levels of other biomarkers such as hs-troponins, hs-CRP will be measured at baseline and after 4 weeks to assess change
Other biomarkers | 6 months
  Levels of other biomarkers such as hs-troponins, hs-CRP will be measured after 6 months.
Symptoms | 4 weeks
  Symptoms will be assessed using a validated, self-administered questionnaire, the Symptom Checklist - Frequency and Severity (SCL). This will be filled out at baseline and 4 weeks to assess change.
Symptoms | 6 months
  Symptoms will be assessed using a validated, self-administered questionnaire, the Symptom Checklist - Frequency and Severity (SCL). This will be filled out at 6 months.
Quality of life in SF-36 | 4 weeks
  The SF-36 (Short Form 36 Health Survey) questionnaire assessing quality of life will be filled out at baseline and 4 weeks to assess change.
Quality of life in SF-36 | 6 months
  The SF-36 questionnaire assessing quality of life will be filled out at 6 months.
Echocardiographic measures - Standard parasternal long axis and three apical views recordings. | 4 weeks
  Will be done in the end expiratory phase with the subjects in supine lateral position. Will be measured at baseline and after 4 weeks to assess change
Echocardiographic measures - Standard parasternal long axis and three apical views recordings. | 6 months
  Will be done in the end expiratory phase with the subjects in supine lateral position. Measured at 6 months.
Echocardiographic measures - Left ventricular dimension, septal and posterior wall thickness. | 4 weeks
  Will be measured as recommended by American Society of Echocardiography. Will be measured at baseline and after 4 weeks to assess change
Echocardiographic measures - Left ventricular dimension, septal and posterior wall thickness. | 6 months
  Will be measured as recommended by American Society of Echocardiography. Measured at 6 months.
Echocardiographic measures - Left ventricular mass. | 4 weeks
  Will be measured as recommended by American Society of Echocardiography. Will be measured at baseline and after 4 weeks to assess change
Echocardiographic measures - Left ventricular mass. | 6 months
  Will be measured as recommended by American Society of Echocardiography. Measured at 6 months.
Echocardiographic measures - Left ventricular and left atrial maximal and minimal volumes. | 4 weeks
  Will be calculated by 2D biplane and 4-chamber and 2D long axis views. (ml/m2). Will be measured at baseline and after 4 weeks to assess change
Echocardiographic measures - Left ventricular and left atrial maximal and minimal volumes. | 6 months
  Will be calculated by 2D biplane and 4-chamber and 2D long axis views. (ml/m2). Measured at 6 months.
Echocardiographic measures - Left ventricular ejection fraction will also be calculated. | 4 weeks
  Using the modified Simpsons rule. Will be measured at baseline and after 4 weeks to assess change
Echocardiographic measures - Left ventricular ejection fraction will also be calculated. | 6 months
  Using the modified Simpsons rule. Measured at 6 months.
Echocardiographic measures - Transmitral flow and pulmonary venous flow. | 4 weeks
  Will be assessed by pulsed Doppler. Tissue Doppler imaging-derived indices will be recorded at the base of the septal and lateral mitral annulus. (cm/s). Will be measured at baseline and after 4 weeks to assess change
Echocardiographic measures - Transmitral flow and pulmonary venous flow. | 6 months
  Will be assessed by pulsed Doppler. Tissue Doppler imaging-derived indices will be recorded at the base of the septal and lateral mitral annulus. (cm/s). Measured at 6 months.
Echocardiographic measures - Global and regional longitudinal left ventricular strain. | 4 weeks
  Will be analysed by a semi-automated speckle tracking technique. Will be measured at baseline and after 4 weeks to assess change
Echocardiographic measures - Global and regional longitudinal left ventricular strain. | 6 months
  Will be analysed by a semi-automated speckle tracking technique.Measured at 6 months.
Echocardiographic measures - Left atrial deformation for assessment of global as well as regional left atrial strain. | 4 weeks
  Will be analysed by a semi-automated speckle tracking technique. Characterizing both reservoir and conduit function. Will be measured at baseline and after 4 weeks to assess change
Echocardiographic measures - Left atrial deformation for assessment of global as well as regional left atrial strain. | 6 months
  Will be analysed by a semi-automated speckle tracking technique. Characterizing both reservoir and conduit function. Measured at 6 months.

OTHER OUTCOMES:
Blood pressure | 4 weeks
  Blood pressure will be measured at baseline and after 4 weeks to assess change
Blood pressure | 6 months
  Blood pressure will be measured after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sara Reinvik Ulimoen, MD PhD, Principal Investigator — Vestre Viken HF Baerum Hospital
Locations (1):
- Vestre Viken Hospital Trust, Baerum Hospital, Rud, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ulimoen SR, Enger S, Pripp AH, Abdelnoor M, Arnesen H, Gjesdal K, Tveit A. Calcium channel blockers improve exercise capacity and reduce N-terminal Pro-B-type natriuretic peptide levels compared with beta-blockers in patients with permanent atrial fibrillation. Eur Heart J. 2014 Feb;35(8):517-24. doi: 10.1093/eurheartj/eht429. Epub 2013 Oct 17. PMID 24135831
- [Background] Ulimoen SR, Enger S, Carlson J, Platonov PG, Pripp AH, Abdelnoor M, Arnesen H, Gjesdal K, Tveit A. Comparison of four single-drug regimens on ventricular rate and arrhythmia-related symptoms in patients with permanent atrial fibrillation. Am J Cardiol. 2013 Jan 15;111(2):225-30. doi: 10.1016/j.amjcard.2012.09.020. Epub 2012 Oct 27. PMID 23111138
- [Background] Go AS, Hylek EM, Phillips KA, Chang Y, Henault LE, Selby JV, Singer DE. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA. 2001 May 9;285(18):2370-5. doi: 10.1001/jama.285.18.2370. PMID 11343485
- [Background] Van Gelder IC, Groenveld HF, Crijns HJ, Tuininga YS, Tijssen JG, Alings AM, Hillege HL, Bergsma-Kadijk JA, Cornel JH, Kamp O, Tukkie R, Bosker HA, Van Veldhuisen DJ, Van den Berg MP; RACE II Investigators. Lenient versus strict rate control in patients with atrial fibrillation. N Engl J Med. 2010 Apr 15;362(15):1363-73. doi: 10.1056/NEJMoa1001337. Epub 2010 Mar 15. PMID 20231232
- [Background] European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery; Camm AJ, Kirchhof P, Lip GY, Schotten U, Savelieva I, Ernst S, Van Gelder IC, Al-Attar N, Hindricks G, Prendergast B, Heidbuchel H, Alfieri O, Angelini A, Atar D, Colonna P, De Caterina R, De Sutter J, Goette A, Gorenek B, Heldal M, Hohloser SH, Kolh P, Le Heuzey JY, Ponikowski P, Rutten FH. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). Eur Heart J. 2010 Oct;31(19):2369-429. doi: 10.1093/eurheartj/ehq278. Epub 2010 Aug 29. No abstract available. PMID 20802247
- [Background] Ulimoen SR, Enger S, Norseth J, Pripp AH, Abdelnoor M, Arnesen H, Gjesdal K, Tveit A. Improved rate control reduces cardiac troponin T levels in permanent atrial fibrillation. Clin Cardiol. 2014 Jul;37(7):422-7. doi: 10.1002/clc.22281. Epub 2014 Apr 3. PMID 24700386
- [Background] Van Gelder IC, Hobbelt AH, Mulder BA, Rienstra M. Rate control in atrial fibrillation: many questions still unanswered. Circulation. 2015 Oct 27;132(17):1597-9. doi: 10.1161/CIRCULATIONAHA.115.018952. Epub 2015 Sep 17. No abstract available. PMID 26384161
- [Derived] Enge K, Ulimoen SR, Enger S, Onarheim S, Olufsen M, Pripp AH, Steinsvik T, Hall C, Hetland M, Tveit A. Effects of diltiazem and metoprolol on levels of high-sensitivity troponin I in patients with permanent atrial fibrillation: a randomized trial. BMC Cardiovasc Disord. 2025 Mar 14;25(1):181. doi: 10.1186/s12872-025-04574-2. PMID 40087560